CLINICAL TRIAL: NCT03048682
Title: Timing of Repeat Voiding Trials After Outpatient Pelvic Floor Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Eric Hurtado, Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FLA 16-123
Record Dates: First submitted 2017-01-26; First posted 2017-02-09 (Estimated); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence,Stress; Surgery
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Voiding Trial (Experimental): All subjects that are discharged home with a Foley catheter will need an in-office repeat voiding trial.
  Subjects in this group will have their repeat voiding trial on post-op day #2, 3, or 4
  Interventions: Device: Foley catheter - Early Voiding Trial
- Late Voiding Trial (Active Comparator): All subjects that are discharged home with a Foley catheter will need an in-office repeat voiding trial.
  Subjects in this group will have their repeat voiding trial on post-op day #7 or after. This is our current practice.
  Interventions: Device: Foley catheter - Late Voiding Trial

INTERVENTIONS:
Device: Foley catheter - Early Voiding Trial — All subjects that are discharged home with a Foley catheter will need an in-office repeat voiding trial.
  Subjects in the Early Voiding group will have their repeat voiding trial on post-op day #2, 3, or 4 will undergo an in-office voiding trial. The experimental group will return for an in-office voiding trial sooner than the active comparator.
  Arms: Early Voiding Trial
Device: Foley catheter - Late Voiding Trial — All subjects that are discharged home with a Foley catheter will need an in-office repeat voiding trial.
  Subjects in the Late Voiding group will have their repeat voiding trial on post-op day #7 or after. This is our current practice
  Arms: Late Voiding Trial

SUMMARY:
This study is a randomized controlled trial designed to assess the rate of failure of voiding trials in the early and late post-operative period within patients who underwent outpatient pelvic floor surgery that failed initial same day voiding trials.

DETAILED DESCRIPTION:
This study would be powered to detect differences in UTIs and Foley catheter re-insertion rates. Assuming a 10% drop-out rate, 100 total subjects should be enrolled in the study.

All patients that meet the appropriate inclusion criteria and are scheduled for outpatient pelvic floor surgery will be considered for the study. Patients will be counseled about the study either in the office during a surgical planning office visit, over a pre-operative telephone call, or in the pre-operative area just prior to surgery. Consents will be signed in the pre-operative area.

After surgery, the patient will be given a standardized voiding trial as per the usual protocol. If the patient is un-successful in emptying her bladder she will be discharged home with an indwelling Foley catheter with antibiotics. On post-operative day (POD) #1 the patient will be re-assessed for meeting eligibility requirements and will be called and randomized to either the early voiding trial group (EVT) or the late voiding trial group (LVT). Subjects in EVT will be scheduled for a repeat VT on POD#2, POD#3, or POD#4, whereas those in LVT will be scheduled for a repeat VT on or after POD#7. Subjects that are unsuccessful in the repeat VT will have a Foley catheter re-inserted and will return for another VT in 5-7 days. Subjects who fail the third VT from either group will have the Foley catheter replaced and will return for another office VT after waiting an additional 5-7 days or will be started on clean intermittent self-catheterization.

Subjects will be monitored for a 6 week period for voiding and urinary symptoms. Urine will be tested via in-office urinalysis at each office visit, including pre-operatively, and will be sent for a urine culture per usual practice based upon abnormal urinalysis results. Urine cultures that grow out a single organism >10,000 CFU will be treated with appropriate antibiotics. In addition, patients will complete quality of life questionnaires at the time of catheter removal, the standard 2 week post-op visit and at 6weeks post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Over 18 years old
* Speak English and are capable of giving informed consent and are able to complete the English patient questionnaire
* Are willing to return to the office for all necessary visits associated with the study
* Had outpatient gynecology pelvic floor surgery for prolapse or stress urinary incontinence
* Failed the voiding trial in the recovery room
* Discharged to home on POD#0

Exclusion Criteria:

* Pre-operative urinary retention as defined as PVR > 200ml
* Prior incontinence surgery
* Passed the voiding trial in the recovery room
* Require prolonged catheterization due to urethral/bladder abnormality (ie vesicovaginal fistula, urethral diverticulum) or intra-op urethral or bladder injury or for intensive post-operative monitoring
* Patients who take any post-operative antibiotics, other than prophylaxis during catheterization, for reasons other than a UTI as diagnosed and prescribed as part of the study
* Patients who take any supplements to prevent UTIs, including but not limited to D-Mannose, Hiprex, or Ellura
* Receive any post-operative vaginal estrogen during the study period
* Have any neurological conditions that may affect bladder function (ie. Multiple sclerosis, spinal cord injuries, etc.)
* Patients with pre-operative narcotic medication use due to chronic pain
* Patients who take any over-active bladder medication within one week of their surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Schachar, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Wake Forest Baptist Health, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
There no plan to make individual participant data available to other researchers

REFERENCES:
- [Background] Alonzo-Sosa JE, Flores-Contreras JT, Paredes-Canul M. [Method for transurethral catheterization for 1-3 days for pelvic floor relaxation in the postoperative period]. Ginecol Obstet Mex. 1997 Nov;65:455-7. Spanish. PMID 9441144
- [Background] Chong C, Kim HS, Suh DH, Jee BC. Risk factors for urinary retention after vaginal hysterectomy for pelvic organ prolapse. Obstet Gynecol Sci. 2016 Mar;59(2):137-43. doi: 10.5468/ogs.2016.59.2.137. Epub 2016 Mar 16. PMID 27004205
- [Background] Ferrante KL, Kim HY, Brubaker L, Wai CY, Norton PA, Kraus SR, Shepherd J, Sirls LT, Nager CW; Urinary Incontinence Treatment Network. Repeat post-op voiding trials: an inconvenient correlate with success. Neurourol Urodyn. 2014 Nov;33(8):1225-8. doi: 10.1002/nau.22489. Epub 2013 Aug 27. PMID 23983149
- [Background] Glavind K, Morup L, Madsen H, Glavind J. A prospective, randomised, controlled trial comparing 3 hour and 24 hour postoperative removal of bladder catheter and vaginal pack following vaginal prolapse surgery. Acta Obstet Gynecol Scand. 2007;86(9):1122-5. doi: 10.1080/00016340701505317. PMID 17712655
- [Background] Hakvoort RA, Elberink R, Vollebregt A, Ploeg T, Emanuel MH. How long should urinary bladder catheterisation be continued after vaginal prolapse surgery? A randomised controlled trial comparing short term versus long term catheterisation after vaginal prolapse surgery. BJOG. 2004 Aug;111(8):828-30. doi: 10.1111/j.1471-0528.2004.00181.x. PMID 15270931
- [Background] Kandadai P, Duenas-Garcia OF, Pilzeck AL, Saini J, Flynn MK, Leung K, Patterson D. A Randomized Controlled Trial of Patient-Controlled Valve Catheter and Indwelling Foley Catheter for Short-term Bladder Drainage. Female Pelvic Med Reconstr Surg. 2016 Mar-Apr;22(2):88-92. doi: 10.1097/SPV.0000000000000249. PMID 26829348
- [Background] Kenton K, Pham T, Mueller E, Brubaker L. Patient preparedness: an important predictor of surgical outcome. Am J Obstet Gynecol. 2007 Dec;197(6):654.e1-6. doi: 10.1016/j.ajog.2007.08.059. PMID 18060968
- [Background] Nicolle LE. Catheter associated urinary tract infections. Antimicrob Resist Infect Control. 2014 Jul 25;3:23. doi: 10.1186/2047-2994-3-23. eCollection 2014. PMID 25075308
- [Background] Ripperda CM, Kowalski JT, Chaudhry ZQ, Mahal AS, Lanzer J, Noor N, Good MM, Hynan LS, Jeppson PC, Rahn DD. Predictors of early postoperative voiding dysfunction and other complications following a midurethral sling. Am J Obstet Gynecol. 2016 Nov;215(5):656.e1-656.e6. doi: 10.1016/j.ajog.2016.06.010. Epub 2016 Jun 16. PMID 27319367
- [Background] Schiotz HA. Comparison of 1 and 3 days' transurethral Foley catheterization after retropubic incontinence surgery. Int Urogynecol J Pelvic Floor Dysfunct. 1996;7(2):98-101. doi: 10.1007/BF01902381. PMID 8798095
- [Background] Schiotz HA, Tanbo TG. Postoperative voiding, bacteriuria and urinary tract infection with Foley catheterization after gynecological surgery. Acta Obstet Gynecol Scand. 2006;85(4):476-81. doi: 10.1080/00016340500409877. PMID 16612711
- [Background] Tan GW, Chan SP, Ho CK. Is transurethral catheterisation the ideal method of bladder drainage? A survey of patient satisfaction with indwelling transurethral urinary catheters. Asian J Surg. 2010 Jan;33(1):31-6. doi: 10.1016/S1015-9584(10)60006-1. PMID 20497880
- [Background] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837
- [Background] Wheeler TL 2nd, Richter HE, Greer WJ, Bowling CB, Redden DT, Varner RE. Predictors of success with postoperative voiding trials after a mid urethral sling procedure. J Urol. 2008 Feb;179(2):600-4. doi: 10.1016/j.juro.2007.09.080. Epub 2007 Dec 21. PMID 18082219

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Voiding Trial: All subjects that are discharged home with a Foley catheter will need an in-office repeat voiding trial.
  Subjects in this group will have their repeat voiding trial on post-op day #2, 3, or 4
  Foley catheter - Early Voiding Trial: All subjects that are discharged home with a Foley catheter will need an in-office repeat voiding trial.
  Subjects in the Early Voiding group will have their repeat voiding trial on post-op day #2, 3, or 4 will undergo an in-office voiding trial. The experimental group will return for an in-office voiding trial sooner than the active comparator.
- Late Voiding Trial: All subjects that are discharged home with a Foley catheter will need an in-office repeat voiding trial.
  Subjects in this group will have their repeat voiding trial on post-op day #7 or after. This is our current practice.
  Foley catheter - Late Voiding Trial: All subjects that are discharged home with a Foley catheter will need an in-office repeat voiding trial.
  Subjects in the Late Voiding group will have their repeat voiding trial on post-op day #7 or after. This is our current practice
Period: Overall Study
Arm/Group | Early Voiding Trial | Late Voiding Trial
Started | 32 | 32
Completed | 30 | 30
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Voiding Trial | Late Voiding Trial | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.06 (12.04) | 65.31 (11.45) | 64.69 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 23 | 26 | 49
  Hispanic | 3 | 5 | 8
  African American | 6 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.24 (6.77) | 26.34 (5.23) | 27.29 (6.07)
Smoking status [Count of Participants; unit: Participants]
  Current | 0 | 0 | 0
  Former | 4 | 5 | 9
  Never | 28 | 27 | 55
Postmenopausal [Count of Participants; unit: Participants] | 28 | 27 | 55
prior hysterectomy [Count of Participants; unit: Participants] | 8 | 9 | 17
POP-Q stage [Count of Participants; unit: Participants] — Subjects are staged clinically using the standard Pelvic Organ Prolapse Quantification system. Increased stage correlates with worsening pelvic organ prolapse.
  Participants
    POP- Q Stage II | 15 | 10 | 25
    POP- Q Stage III | 15 | 21 | 36
    POP-Q Stage IV | 2 | 1 | 3
pre-operative post void residual [Mean (Standard Deviation); unit: ml] | 38.84 (30.11) | 38.94 (39.62) | 38.89 (34.90)
Urodynamic diagnosed incontinence [Count of Participants; unit: Participants] — Population: Not all subjects underwent urodynamic testing.
  Participants
    number analyzed (Participants) | 28 | 29 | 57
    None | 14 | 14 | 28
    SUI | 11 | 9 | 20
    ISD | 2 | 3 | 5
    DO | 1 | 3 | 4
Concurrent vaginal hysterectomy [Count of Participants; unit: Participants] | 21 | 11 | 32
Apical Suspension [Count of Participants; unit: Participants] | 25 | 27 | 52
Type of Apical Suspension [Count of Participants; unit: Participants] — Population: Not all subjects underwent an apical suspension
  Participants
    number analyzed (Participants) | 25 | 27 | 52
    Sacrospinous Fixation | 10 | 14 | 24
    Uterosacral Suspension | 15 | 13 | 28
Anterior Colporrhaphy [Count of Participants; unit: Participants] | 24 | 27 | 51
Posterior Colporrhaphy [Count of Participants; unit: Participants] | 30 | 32 | 62
Midurethral Sling [Count of Participants; unit: Participants] | 18 | 14 | 32
Vaginal Pack Used [Count of Participants; unit: Participants] | 15 | 13 | 28
Intra-operative Urine Dye [Count of Participants; unit: Participants]
  None | 18 | 23 | 41
  Fluorescein | 7 | 3 | 10
  Indigo Carmine | 5 | 5 | 10
  Phenazopyridine | 2 | 1 | 3
Intra-operative use of Furosemide [Count of Participants; unit: Participants] | 4 | 5 | 9
Anesthesia [Count of Participants; unit: Participants]
  General | 31 | 32 | 63
  Spinal | 1 | 0 | 1
Total Morphine Dose Equivalents [Mean (Standard Deviation); unit: morphine dose equivalents] | 21.45 (11.85) | 18.67 (8.72) | 20.06 (10.41)

OUTCOME MEASURES:

1. Primary Outcome: Failed Office Voiding Trials
Description: Determine the rates of failed voiding trials in each of the two groups
Time Frame: within 8 days of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Early Voiding Trial | Late Voiding Trial
Number analyzed (Participants) | 30 | 30
Participants | 7 | 1

2. Secondary Outcome: Urinary Tract Infections
Description: Determine the rates of urinary tract infections in each of the two groups
Time Frame: within 6 weeks of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Early Voiding Trial | Late Voiding Trial
Number analyzed (Participants) | 30 | 30
Participants | 7 | 2

3. Secondary Outcome: Rate of Bother From Urinary Catheter
Description: Determine the rates of patient satisfaction in each of the two groups using a Likert scale (1= very bothersome; 5= Not bothersome at all)
Time Frame: within 6 weeks of surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Early Voiding Trial | Late Voiding Trial
Number analyzed (Participants) | 30 | 30
score on a scale | 3 [1 to 3.5] | 2 [1 to 3]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Early Voiding Trial | Late Voiding Trial
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03048682/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-12-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT03048682/SAP_001.pdf